CLINICAL TRIAL: NCT05331521
Title: Improvement of Functional Outcome for Patients With Newly Diagnosed Grade 2 or 3 Glioma With Co-deletion of 1p/19q - IMPROVE CODEL: the NOA-18 Trial
Brief Title: A Clinical Study to Improve Brain Function and Quality of Life of Patients With Newly Diagnosed Brain Tumors (Gliomas).
Acronym: ImproveCodel
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Universitätsmedizin Mannheim (Other); Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Prof. Dr. Wolfgang Wick, Medical Director of Neurology, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NOA-18; 2018-005027-16 (EudraCT Number); 2024-510616-73-00 (EU CTIS Number)
Record Dates: First submitted 2022-03-15; First posted 2022-04-15 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Oligodendroglioma
Keywords: Radiotherapy; Chemotherapy; Temozolomide
MeSH Terms: conditions — Oligodendroglioma | interventions — Lomustine; Temozolomide; Procarbazine; Vincristine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RT PCV (Active Comparator): Radiotherapy (RT) for over approximately 5-6 weeks:
  * at 50.4/54 Gy in 1.8 Gy fractions for grade 2 and
  * at 59.4 Gy in 1.8 Gy fractions for grade 3 gliomas
  PCV cycles are 6 weeks long and given as:
  * Day 1: Lomustine (CCNU) at 110 mg/m2 body surface orally,
  * Days 8/29: Vincristine 1.4 mg/m2 i.v. (capped at 2 mg),
  * Days 8-21: Procarbazine 60 mg/m2 orally (capped at 100 mg).
  Interventions: Drug: PCV; Radiation: RT
- CETEG (Experimental): Six 42-day cycles of lomustine plus temozolomide according to the commonly used regimen:
  * Day 1: Lomustine (CCNU) at 100 mg/m2
  * Days 2-6: Temozolomide at 100 mg/m2 (cycles 1) and in 50 mg/m2 steps to 200 mg/m2 from cycle 2 on dependent on hematological toxicity
  Interventions: Drug: CETEG

INTERVENTIONS:
Drug: CETEG — At progression, patients without prior radiotherapy will undergo radiotherapy and PCV as an adjunct chemotherapy if bone marrow reserve allows in the experimental arm.
  Other Names: Lomustine (CCNU) and Temozolomide
  Arms: CETEG
Drug: PCV — In the comparator arm there is the option for second radiotherapy or even reuse of the full radiochemotherapy regimen as it had been given at diagnosis (BIC).
  Other Names: Procarbazine, Lomustine and Vincristine
  Arms: RT PCV
Radiation: RT — Radiotherapy at 50.4/54 Gy in 1.8 Gy fractions for grade 2 and 59.4 Gy in 1.8 Gy fractions for grade 3 gliomas
  Other Names: Radiotherapy
  Arms: RT PCV

SUMMARY:
Oligodendrogliomas in the novel edition of the Central Nervous System (CNS) World Health Organization (WHO) classification are now molecularly defined by isocitrate dehydrogenase (IDH)1 or IDH2 mutations and 1p/19q co-deletion. The prognosis of these molecularly defined tumors is to be determined in new series since survival data from older histology-based studies and population-based registries are confounded by the inclusion of 20-70% not molecularly matching subsets. Also, the optimal treatment is a matter of ongoing investigations. An extensive, but safe surgery is associated with improved outcome as is the addition of chemotherapy with procarbazine, CCNU (lomustine), and vincristine (PCV) to the partial brain radiotherapy (RT). However, the exact timing of postsurgical therapy especially for tumors of the WHO grade 2 and acknowledging some variability in grading as well as the choice of chemotherapy, temozolomide instead of PCV (CODEL: NCT00887146 randomizing CNS WHO grade 2 and 3 oligodendrogliomas to chemoradiation(CHRT)therapy with PCV or with temozolomide) or the need for primary radiotherapy RT are subjects of clinical studies (POLCA: NCT02444000 randomizing patients with newly diagnosed CNS WHO grade 3 oligodendrogliomas to standard CHRT with PCV or PCV alone). Given the young age of patients with CNS WHO grade 2 and 3 oligodendrogliomas and the relevant risk of neurocognitive, functional and quality-of-life impairment with the current aggressive standard of care treatment, chemoradiation with PCV, of the tumor located in the brain optimizing care is the major challenge.

NOA-18/IMPROVE CODEL aims at improving qualified overall survival (qOS) for adult patients with CNS WHO grade 2 and 3 oligodendrogliomas by randomizing between standard chemoradiation with up to six six-weekly cycles with PCV and six six-weekly cycles with lomustine and temozolomide (CETEG), thereby delaying radiotherapy (RT) and adding the chemoradiotherapy (CHRT) concept at progression after initial radiation-free chemotherapy, allowing for an effective salvage treatment and delaying potentially deleterious side effects. QOS represents a new concept and is defined as OS without functional and/or cognitive and/or quality of life (QOL) deterioration regardless whether tumor progression or toxicity is the main cause.

DETAILED DESCRIPTION:
The primary objective of the NOA-18/IMPROVE CODEL trial is to show superiority of an initial CETEG treatment followed by partial brain radiotherapy (RT) plus PCV (RT-PCV) at progression over partial brain radiotherapy (RT) followed by procarbazine, lomustine and vincristine (PCV) chemotherapy (RT-PCV) and best investigators choice (BIC) at progression for sustained qOS. An event with respect to a sustained qOS is then defined as a functional and/or cognitive deterioration on two consecutive study visits with an interval of 3 months, tolerating a deviation of at most 1 month. Assessments are done with 3-monthly MRI, assessment of the NANO (Neurologic assessment in neuro-oncology) scale, HRQoL, and KPS (Karnofsky performance status) and annually cognitive testing. Secondary objectives are evaluation and comparison of the two groups regarding secondary endpoints (short-term qOS, PFS, OS, complete and partial response rate). The trial is planned to be conducted at 21 NOA (Neurooncology Working Party of the German Cancer Society) study sites in Germany.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed, newly diagnosed CNS WHO grade 2 or 3 glioma.
2. Tumor carries an isocitrate dehydrogenase (IDH) mutation (determined by immunohistochemistry (IHC) and/or deoxyribonucleic acid (DNA) sequencing).
3. Tumor is co-deleted for 1p/19q (determined by copy number variations, fluorescence in situ hybridization (FISH), multiplex ligation-dependent probe amplification (MLPA) or other appropriate methods).
4. Biopsy (with sufficient tissue for molecular pathology) or resection.
5. Age: ≥18 years.
6. Karnofsky Performance status (KPI) ≥60%.
7. Life expectancy >6 months.
8. Availability of formalin-fixed paraffin-embedded (FFPE) or fresh-frozen tissue and ethylenediamine tetraacetic acid (EDTA) blood for biomarker research.
9. Standard magnetic resonance imaging (MRI) ≤ 72 h post-surgery according to the present national and international guidelines.
10. Craniotomy or intracranial biopsy site must be adequately healed.
11. ≥ 2 weeks and ≤ 3 months from surgery without any interim radio- or chemotherapy or experimental intervention.
12. Willing and able to comply with regular neurocognitive and health-related quality of life tests/questionnaires.
13. Indication for postsurgical cytostatic/-toxic therapy.
14. Written Informed consent.
15. Female patients with reproductive potential have a negative pregnancy test (serum or urine) day -6 until day 0 of screening (and 3 days prior to first IMP-intake or RT). Female patients are surgically sterile or agree to use adequate contraception during the period of therapy and 7 months after the end of study treatment, or women have been postmenopausal for at least 2 years.
16. Male patients are willing to use contraception

Exclusion Criteria:

1. Participation in other ongoing interventional clinical trials.
2. Inability to undergo MRI.
3. Abnormal (≥ Grade 2 CTCAE v5.0 laboratory values for hematology (Hb, WBC, neutrophils, or platelets), liver (serum bilirubin, ALT, or AST) or renal function (serum creatinine).
4. Clinically active tuberculosis; known HIV infection or active Hepatitis B (HBV) or Hepatitis C (HCV) infection, or active infections requiring oral or intravenous antibiotics or that can cause a severe disease and pose a severe danger to lab personnel working on patients' blood or tissue (e.g. rabies).
5. Any prior anti-cancer therapy or co-administration of anti-cancer therapies other than those administered/allowed in this study. History of low-grade glioma that did not require prior treatment with chemotherapy or radiotherapy is not an exclusion criterion.
6. Immunosuppression, not related to prior treatment for malignancy.
7. History of other malignancies (except for adequately treated basal or squamous cell carcinoma or carcinoma in situ) within the last 5 years unless the patient has been disease-free for 5 years.
8. Any clinically significant concomitant disease (including hereditary fructose intolerance) or condition that could interfere with, or for which the treatment might interfere with, the conduct of the study or the absorption of oral medications or that would, in the opinion of the Principal Investigator, pose an unacceptable risk to the patient in this study.
9. Any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol requirements and/or follow-up procedures; those conditions should be discussed with the patient before trial entry.
10. Pregnancy or breastfeeding.
11. History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product. (E.g.: In the discretion of the investigator patients are allowed to take part in the study even if they suffer from celiac disease: Cecenu contains very small amounts of gluten (from wheat starch). It is considered gluten-free and is tolerated by patients suffering from celiac disease. One capsule contains no more than 4 micrograms of Gluten.)
12. QTc time prolongation >500 ms.
13. Patients under restricted medication for procarbazine, lomustine, vincristine and temozolomide.
14. Liver disease characterized by:

    1. ALT or AST (≥ Grade 2 CTCAE v5.0) confirmed on two consecutive measurements OR
    2. Impaired excretory function (e.g., hyperbilirubinemia) or synthetic function or other conditions of decompensated liver disease such as coagulopathy, hepatic encephalopathy, hypoalbuminemia, ascites, and bleeding from esophageal varices (≥ Grade 2 CTCAE v5.0) OR
    3. Acute viral or active autoimmune, alcoholic, or other types of acute hepatitis.
15. Known uncorrected coagulopathy, platelet disorder, or history of non-drug induced thrombocytopenia.
16. History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis; autoimmune-related hypothyroidism (patients on a stable dose of thyroid replacement hormone are eligible for this study) and type I diabetes mellitus (patients on a stable dose of insulin regimen are eligible for this study).
17. Vaccination with life vaccines during treatment and 4 weeks before start of treatment.
18. Existing neuromuscular diseases, especially neural muscular atrophy with segmental demyelination (demyelinising form of Charcot-Marie-Tooth syndrome).
19. Chronic constipation and subileus.
20. Combination treatment with mitomycin (risk of a pronounced bronchospasm and acute shortness of breath).
21. Hypersensitivity to dacarbazine (DTIC).
22. Patients with hereditary galactose intolerance, complete lactase deficiency or glucose-galactose malabsorption (Temodal contains Lactose).
23. Patients with clinical wheat allergy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Estimated)
Dates: Start 2021-04-07 (Actual); Primary Completion 2033-03-31 (Estimated); Study Completion 2033-03-31 (Estimated)

PRIMARY OUTCOMES:
Qualified overall survival (qOS) | Counted as event starting 12 months (365 days) after randomization on 2 consecutive study visits with an interval of 3 months (90 days) till the end of follow up at 120 months or date of death from any cause, whatever occurs first.
  The primary efficacy endpoint is the overall survival without functional and/or cognitive and/or quality of life deterioration over a period of 90 days, coined qualified overall survival (qOS).
Short-term qOS deterioration in NeuroCogFX® | Counted as event starting 12 months (365 days) after randomization on 2 consecutive study visits with an interval of 3 months (90 days) till the end of follow up at 120 months or date of death from any cause, whatever occurs first.
  The primary efficacy endpoint is overall survival without functional and/or cognitive and/or quality of life deterioration over a period of 90 days, coined qualified overall survival (qOS). Short-term qOS is defined as detriment of ≥ 1.5 standard deviations below the normative mean (i.e. percentile rank ≤ 6.68) in two or more NeuroCog FX® subtests AND Related to baseline: 90%-confidence intervals of NeuroCog FX® subtests indicate a clinically and statistically meaningful individual change (i.e. deterioration) in two or more NeuroCog FX® subtest raw scores
Short-term qOS deterioration in KPI | Counted as event starting 12 months (365 days) after randomization on 2 consecutive study visits with an interval of 3 months (90 days) till the end of follow up at 120 months or date of death from any cause, whatever occurs first.
  The primary efficacy endpoint is overall survival without functional and/or cognitive and/or quality of life deterioration over a period of 90 days, coined qualified overall survival (qOS). Short-term qOS is defined as a decrease in the KPI from 100 or 90 to 70 or less, a decrease in KPI of at least 20 from 80 or less, or a decrease in KPI from any baseline to 50 or less. Fulfilment of one of these criteria is considered neurological deterioration unless attributable to comorbid events or changes in corticosteroid dose.
Short-term qOS deterioration in HrQoL | Counted as event starting 12 months (365 days) after randomization on 2 consecutive study visits with an interval of 3 months (90 days) till the end of follow up at 120 months or date of death from any cause, whatever occurs first.
  The primary efficacy endpoint is overall survival without functional and/or cognitive and/or quality of life deterioration over a period of 90 days, coined qualified overall survival (qOS). Short-term qOS is defined as a worsening of at least 10 points, which is the minimal clinically relevant difference, in at least one of the five selected domains of the HrQoL (global health status (GHS), physical functioning (PF), social functioning (SF), determined in the QLQ-C30 with higher scores indicate better HRQoL; communication deficits (CD) & motor dysfunction (MD) determined by QLQ-BN20 with lower scores indicate better HRQoL).
Short-term qOS deterioration in NANO scale | Counted as event starting 12 months (365 days) after randomization on 2 consecutive study visits with an interval of 3 months (90 days) till the end of follow up at 120 months or date of death from any cause, whatever occurs first.
  The primary efficacy endpoint is overall survival without functional and/or cognitive and/or quality of life deterioration over a period of 90 days, coined qualified overall survival (qOS). Short-term qOS is defined as a decline in the NANO scale defined as a ≥2 level worsening from baseline within ≥1 domain or worsening to the highest score within ≥1 domain that is felt to be related to underlying tumor progression and not attributable to a comorbid event or change in concurrent medication.
Short-term qOS deterioration due to death | From start of randomization until death from any cause till the end of follow up at 120 months.
  Death due to any cause.

SECONDARY OUTCOMES:
Short-term qOS | From 3 months after start of treatment, every 3 months till the end of follow up at 120 months or date of death from any cause, whatever occurs first.
  Defined qOS defined as qOS as described above, but neglecting the subsequent time interval of 3 months (90 days).
Overall survival (OS) | From start of randomization until death from any cause till the end of follow up at 120 months.
  Defined as the time from randomization until death due to any cause.
Progression-free survival (PFS) | From randomization until the day of first documentation of clinical or radiographic tumor progression or death of any cause till the end of follow up at 120 months or date of death from any cause, whatever occurs first.
  Defined as the time from randomization to the day of first documentation of clinical or radiographic tumor progression or death of any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Wick, Prof. Dr., Principal Investigator — University Hospital Heidelberg
Locations (19):
- Germany (19):
  - University Hospital Heidelberg, Department of Neurooncology, Heidelberg, Baden-Wurttemberg
  - Charité, University Medicine Berlin, Neurosurgery, Berlin
  - Knappschaftskrankenhaus Bochum GmbH, Neurology Clinic, Bochum
  - University Hospital Bonn, Neurology Clinic, Bonn
  - Chemnitz Hospital, Neurosurgery, Chemnitz
  - University Hospital Cologne, Neurosurgery, Cologne
  - University Hospital Duesseldorf, Neurooncology, Düsseldorf
  - University Hospital Frankfurt, Neurooncology, Frankfurt
  - University Hospital Göttingen, Neurosurgery, Göttingen
  - University Hospital Saarland, Neurosurgery, Homburg
  - University Hospital of Jena, Neurosurgery, Jena
  - University Hospital Leipzig, Radiation Therapy, Leipzig
  - University Hospital Mannheim, Neurology Clinic, Mannheim
  - University Clinic Muehlenkreis, Minden, Minden
  - University Hospital rechts der Isar, Radiation Oncology, Munich
  - University Hospital Regensburg, Neurology Clinic, Regensburg
  - Helios Hospital Schwerin, Neurosurgery, Schwerin
  - University Hospital Tuebingen, Neurooncology, Tübingen
  - University Hospital Wuerzburg, Neurosurgery, Würzburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Louis DN, Perry A, Wesseling P, Brat DJ, Cree IA, Figarella-Branger D, Hawkins C, Ng HK, Pfister SM, Reifenberger G, Soffietti R, von Deimling A, Ellison DW. The 2021 WHO Classification of Tumors of the Central Nervous System: a summary. Neuro Oncol. 2021 Aug 2;23(8):1231-1251. doi: 10.1093/neuonc/noab106. PMID 34185076
- [Background] Weller M, van den Bent M, Preusser M, Le Rhun E, Tonn JC, Minniti G, Bendszus M, Balana C, Chinot O, Dirven L, French P, Hegi ME, Jakola AS, Platten M, Roth P, Ruda R, Short S, Smits M, Taphoorn MJB, von Deimling A, Westphal M, Soffietti R, Reifenberger G, Wick W. EANO guidelines on the diagnosis and treatment of diffuse gliomas of adulthood. Nat Rev Clin Oncol. 2021 Mar;18(3):170-186. doi: 10.1038/s41571-020-00447-z. Epub 2020 Dec 8. PMID 33293629
- [Background] Fliessbach K, Rogowski S, Hoppe C, Sabel M, Goeppert M, Helmstaedter C, Calabrese P, Schackert G, Tonn JC, Simon M, Schlegel U. Computer-based assessment of cognitive functions in brain tumor patients. J Neurooncol. 2010 Dec;100(3):427-37. doi: 10.1007/s11060-010-0194-9. Epub 2010 May 7. PMID 20449630
- [Background] Hoffermann M, Bruckmann L, Mahdy Ali K, Zaar K, Avian A, von Campe G. Pre- and postoperative neurocognitive deficits in brain tumor patients assessed by a computer based screening test. J Clin Neurosci. 2017 Feb;36:31-36. doi: 10.1016/j.jocn.2016.10.030. Epub 2016 Nov 9. PMID 27836394
- [Background] Taphoorn MJ, Henriksson R, Bottomley A, Cloughesy T, Wick W, Mason WP, Saran F, Nishikawa R, Hilton M, Theodore-Oklota C, Ravelo A, Chinot OL. Health-Related Quality of Life in a Randomized Phase III Study of Bevacizumab, Temozolomide, and Radiotherapy in Newly Diagnosed Glioblastoma. J Clin Oncol. 2015 Jul 1;33(19):2166-75. doi: 10.1200/JCO.2014.60.3217. Epub 2015 May 26. PMID 26014298
- [Background] Nayak L, DeAngelis LM, Brandes AA, Peereboom DM, Galanis E, Lin NU, Soffietti R, Macdonald DR, Chamberlain M, Perry J, Jaeckle K, Mehta M, Stupp R, Muzikansky A, Pentsova E, Cloughesy T, Iwamoto FM, Tonn JC, Vogelbaum MA, Wen PY, van den Bent MJ, Reardon DA. The Neurologic Assessment in Neuro-Oncology (NANO) scale: a tool to assess neurologic function for integration into the Response Assessment in Neuro-Oncology (RANO) criteria. Neuro Oncol. 2017 May 1;19(5):625-635. doi: 10.1093/neuonc/nox029. PMID 28453751
- [Background] Wen PY, Macdonald DR, Reardon DA, Cloughesy TF, Sorensen AG, Galanis E, Degroot J, Wick W, Gilbert MR, Lassman AB, Tsien C, Mikkelsen T, Wong ET, Chamberlain MC, Stupp R, Lamborn KR, Vogelbaum MA, van den Bent MJ, Chang SM. Updated response assessment criteria for high-grade gliomas: response assessment in neuro-oncology working group. J Clin Oncol. 2010 Apr 10;28(11):1963-72. doi: 10.1200/JCO.2009.26.3541. Epub 2010 Mar 15. PMID 20231676
- [Background] Wick W, Roth P, Hartmann C, Hau P, Nakamura M, Stockhammer F, Sabel MC, Wick A, Koeppen S, Ketter R, Vajkoczy P, Eyupoglu I, Kalff R, Pietsch T, Happold C, Galldiks N, Schmidt-Graf F, Bamberg M, Reifenberger G, Platten M, von Deimling A, Meisner C, Wiestler B, Weller M; Neurooncology Working Group (NOA) of the German Cancer Society. Long-term analysis of the NOA-04 randomized phase III trial of sequential radiochemotherapy of anaplastic glioma with PCV or temozolomide. Neuro Oncol. 2016 Nov;18(11):1529-1537. doi: 10.1093/neuonc/now133. Epub 2016 Jul 1. PMID 27370396
- [Derived] Wick A, Sander A, Koch M, Bendszus M, Combs S, Haut T, Dormann A, Walter S, Pertz M, Merkle-Lock J, Selkrig N, Limprecht R, Baumann L, Kieser M, Sahm F, Schlegel U, Winkler F, Platten M, Wick W, Kessler T. Improvement of functional outcome for patients with newly diagnosed grade 2 or 3 gliomas with co-deletion of 1p/19q - IMPROVE CODEL: the NOA-18 trial. BMC Cancer. 2022 Jun 13;22(1):645. doi: 10.1186/s12885-022-09720-z. PMID 35692047